CLINICAL TRIAL: NCT06989060
Title: Assessment of Nutritional Status and Detection of Nutritional Deficiencies in Children With Down Syndrome
Brief Title: Nutritional Status in Children With Down Syndrome
Acronym: DS
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Esraa Gamal Gomaa, Principal Investigator, Assiut University
Other Study IDs: nutritional status in DS
Record Dates: First submitted 2025-04-01; First posted 2025-05-25 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Down Syndrome
MeSH Terms: conditions — Down Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
To evaluate the nutritional status of children with Down's syndrome and to determine the prevalence of nutritional deficiencies among those children.

To discuss factors associated with their nutritional status, such as dietary habits and comorbid health conditions.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of children with Down's syndrome Age between 2- 5 years of both sexes

Exclusion Criteria:

Children diagnosed with any other chronic illness or any other medical problem

Ages: 2 Years to 5 Years | Sex: All
Age Groups: Child
Study Population: Children diagnosed with Down's syndrome Age between 2- 5 years of both sexes
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Weight | Baseline
  Body weight of children with Down syndrome will be measured in kilograms using a calibrated scale by trained personnel.
Height | Baseline
  Height of children with Down syndrome will be measured in centimeters using a calibrated stadiometer by trained personnel.
Body Mass Index (BMI) | Baseline
  BMI will be calculated using the formula: weight (kg) divided by height in meters squared (m²). Nutritional status will be classified based on WHO Child Growth Standards (underweight, normal weight, overweight, etc.).

CONTACTS AND LOCATIONS:
Overall Officials: Osama M Asheer, professor of pediatrics, Principal Investigator — assiut university child hospital
Locations (1):
- Assiut university child hospital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No